CLINICAL TRIAL: NCT03411551
Title: Efficacy of Ultrasound-guided Peripheral Nerve Block Versus Forearm Bier's Block in Patients Undergoing Carpal Tunnel Release: A Randomized Controlled Trial
Brief Title: Ultrasound-guided Peripheral Nerve Block Versus Forearm Bier's Block in Patients Undergoing Carpal Tunnel Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Principal Investigator, Anesthesiologist, MD, PhD, Jessa Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17.118/ANESTH17.03
Record Dates: First submitted 2018-01-11; First posted 2018-01-26 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Carpal Tunnel Syndrome; Anesthesia, Local
Keywords: Intravenous anesthesia; Nerve Block; Regional anesthesia
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Anesthesia, Conduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forearm Bier's block (Active Comparator): Forearm intravenous regional anesthesia (Bier's block)
  Interventions: Procedure: regional anesthesia
- Peripheral Nerve Block (Experimental): Ultrasound-guided peripheral nerve block (regional anesthesia)
  Interventions: Procedure: regional anesthesia

INTERVENTIONS:
Procedure: regional anesthesia — The analgesic effectivity of the forearm intravenous regional anesthesia and the ultrasound-guided peripheral nerve block will be investigated in patients undergoing carpal tunnel release

SUMMARY:
By means of an observer-blinded, randomized controlled trial, the analgesic efficacy of the forearm intravenous regional anesthesia and the ultrasound guided peripheral nerve block will be investigated in patients undergoing carpal tunnel release. The hypothesis is that the ultrasound-guided peripheral nerve block is superior compared to the forearm intravenous regional anesthesia with respect to the analgesic efficacy.

Furthermore, pre-, intra-, and post-operative pain will be investigated at several time points as well as general patient satisfaction and satisfaction of the surgeon regarding the procedures.

DETAILED DESCRIPTION:
Introduction:

In Belgium, several ways of anesthesia are used to perform hand surgery, being general anesthesia, intravenous regional anesthesia as well as locoregional anesthesia. Locoregional anesthesia and intravenous regional anesthesia are often performed since patients can be discharged from the hospital more rapidly. A forearm intravenous regional anesthesia (IVRA; mini-Bier's block) is an effective and safe technique to perform hand surgery, especially since the dose of the used anesthetic is reduced compared to a regular upper arm Bier's block, leading to a reduced risk of local anesthetic toxicity. An ultrasound-guided distal peripheral nerve block is often used for hand surgery, in which the nervus medianus and the nervus ulnaris can be affected locally. Research showed that this technique is associated with a reduced surgical procedure time when compared to intravenous regional anesthesia (1). In the Jessa Hospital, a carpal tunnel release is often performed using the forearm intravenous regional anesthesia. However, to date, the analeptic effectivity of the forearm intravenous regional anesthesia has not been compared to the distal peripheral nerve block.

Outcome measures:

The primary aim of this study is to compare the analgesic effectivity of the forearm intravenous regional anesthesia versus the ultrasound-guided distal peripheral nerve block. Our hypothesis is that the latter technique is superior. A blinded surgeon will determine the analgesic effectivity of these techniques (graded as "complete" or "incomplete") and divide the effectivity in 4 grades. Grade 1 and grade 2 are considered "complete" blockade, while grade 3 and grade 4 are considered "incomplete" blockade. Grade 1: complete motor and sensory blockade, grade 2: partial motor blockade but no pain or deep pressure sensitivity, grade 3: partial motor blockade with mild pain requiring rescue local or opioid analgesia, grade 4: incomplete motor- and sensory blockade requiring sedation/conversion to general anesthesia). Secondary study outcomes are patient's pre-, intra-, and post-operative pain scores at several time points, measured via an 11-point Numeric Rating Scale (NRS) in which number 0 means "no pain at all", number 5 means "moderate pain" and number 10 means "worst possible pain". General patient satisfaction as well as satisfaction of the surgeon regarding the used technique will be measured via a 7-point Likert Scale, in which number 1 means "extremely dissatisfied" and number 7 means "extremely satisfied". Furthermore, the time spend in the operating room, the time of surgical procedure and the use of post-operative medication use will be recorded as well.

Design:

In this monocentric, investigator-initiated, observer-blinded, prospective, randomized controlled trial, 2 groups of patients that will undergo carpal tunnel release surgery will be compared. This study will be performed according to the Declaration of Helsinki and will be approved by the Ethical Committee of the Jessa Hospital before the start of the study. A written informed consent will be obtained before participation in the study. Randomization will be performed using a computer-generated random allocation sequence, created by the study statistician. Allocation numbers will be sealed in opaque envelopes, which will be opened in sequence by an independent anaesthesiologist who is not involved in the assessment of outcomes.

Study Procedures:

The patient will first receive information about this study during the consultation with the surgeon. After having ample amount of time to consider participation and before the start of the study, written informed consent will be obtained. Afterwards, the patient will be randomized to one of the 2 study groups. All anesthesia techniques will be performed by only 2 anaesthesiologists, to reduce the inter-individual difference in anaesthesia. All patients will receive an intravenous catheter, supplementary oxygen and standard monitoring (non-invasive blood pressure, electrocardiogram and saturation measurements).

Forearm intravenous regional anesthesia:

An intravenous catheter will be placed in the dorsal vein of the hand that will undergo surgery. Also, a tourniquet will be placed on the forearm, after which the anesthetic can be administered via the dorsal vein catether (25ml linisol 0.5%).

Distal peripheral nerve block:

For the distal peripheral nerve block, a General Electric LOGIQe device and a 12 MHz lineair echotransducer with a foot of 4 cm will be used to locate the nervus medianus and the nervus ulnaris. In total, 10ml linisol 2% will be used to affect the nerves (3ml linisol 2% around the nervus medianus, 3ml linisol 2% around the nervus ulnaris and 4ml linisol 2% around the peripheral distal nerves).

The surgeon and the researcher will be blinded for the used type of anaesthesia. To reduce a possible deblinding, all patients receive a catheter in the dorsal vein of the hand that will undergo surgery and all patients will receive disinfection on the specific locations on the arm where the ultrasound-guided peripheral nerve block would be performed. In that way, both surgeon and researcher are blinded. Before the start of the surgery, the surgeon will assess the quality of the block (primary outcome) in the nervus ulnaris and nervus medianus, using a forceps. The quality of the block will be graded "complete" (grade 1 and grade 2) or "incomplete" (grade 3 or grade 4). In case of grade 1 or grade 2, the surgical procedure can start. In case of grade 3, the blockade will be enhanced (local anesthetic for peripheral nerve block or intravenous opioid administration (alfentanil or sufentanil) for IVRA). In case of grade 4, sedation/conversion to general anesthesia will be performed. Per-operative paracetamol administration 15mg/kg (max 1gram) and taradyl 0.5mg/kg (max 30mg) will be supplied (except when there are contraindications). All patients (both distal peripheral nerve block and IVRA) will receive dexamethasone 0.1mg/kg (max 5mg) (except when there are contraindications) due to the positive effect of dexamethasone on the extension of the locoregional anesthesia and the prevention of post-operative nausea and vomiting. All secondary outcome measures will be investigated by the blinded researcher via questioning the patient's pain scores (measured via an Numeric Rating Scale) at several time points before, during and after surgery, and the satisfaction of both patient and surgeon (measured via a 7-point Likert Scale). Post-operative pain medication in the hospital includes paracetamol 15mg/kg (max 1gr) 1x/6h and taradyl 0.5mg/kg (max 30mg) 1x/8h, while contramal serves as rescue medication. Post-operative pain medication at home includes paracetamol 15mg/kg (max 1gr) 1x/6h or ibuprofen 600mg 1x/8h whenever necessary. On day 1 after surgery, the patient will be contacted via telephone by the researcher who will question the use of post-operative pain medication, as well as NRS pain scores and patient satisfaction.

Statistical analysis:

Sample size was determined for the primary study outcome with the aim to reject the superiority of the distal peripheral nerve block compared to forearm intravenous regional anesthesia. Based on a retrospective analysis of unpublished data from our hospital, we assume that 75% of patients will have a complete block (grade 1 or2) after a forearm IVRA. Based on a previous study, we assume that 95% of patients will have a complete block (grade 1 or 2) after a distal peripheral nerve block (2). By using a binary outcome, we determined the sample size for each group to be 47 (α=0.05, power=0.80). To account for a possible 6% drop-out rate, the sample size was increased to 50 patients per group. Descriptive statistics will be presented as frequencies and percentages of the total amount of patients for categorical variables, while numerical variables will be presented as mean ± SD. Group comparison will be performed using Chi-square test (or a Fisher's Exact test when necessary) for frequencies. Depending on normality, a Mann-Witney U test or a Student's t-test will be used and a Mixed-model analysis will be used to correct for the multiple measurements of the Numerical Rating Scale (NRS) for pain scores. An average difference of 1.3 points or more on the NRS pain score is considered clinical relevant. A p-value <0.05 is considered statistical significant, while p<0.10 is considered a tendency.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 years of age
* American Society of Anesthesiology (ASA) physical status classification: 1-3
* Patients planned to undergo carpal tunnel release via regional anesthesia (intravenous regional anesthesia or ultra-sound guided peripheral nerve block)

Exclusion Criteria:

* Bilateral surgery
* BMI ≥ 40 kg/m2
* Infection in the area of the peripheral nerve block injection site
* History of neurological conditions
* Chronic pain symptoms
* Concomitant use of Opioids in the last 3 months
* Diabetes mellitus type-1 (insulin dependent diabetes mellitus)
* Diabetes mellitus with organ damage
* Oversensitivity to local anesthesia
* Blood clotting disorder
* History of any surgical procedure in the arm that needs to be operated
* Inability to understand and adhere to the study design

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Analgesic effectivity | Intraoperative
  This study wants to evaluate and compare the analgesic effectivity of the intravenous regional anesthesia (IVRA; mini-Bier's block) and the ultrasound-guided peripheral nerve block. The blinded surgeon will assess the analgesic effectivity and grade it as either complete (grade 1 and grade 2) or incomplete (grade 3 and grade 4). Grade 1 is defined as complete motor and sensory blockade; grade 2 is defined as partial motor blockade with no pain or deep pressure sensitivity. Grade 3 is defined as partial motor blockade with mild pain and the need for rescue local or opioid analgesia. Grade 4 is defined as incomplete motor and sensory blockade requiring sedation/conversion to general anesthesia.

SECONDARY OUTCOMES:
Pre operative pain | Start of anesthesia technique
  Pain score at start of anesthesia technique will be assessed via a Numerical Rating Scale (NRS). This scale is ranged (0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10) in which 0 stand for "no pain at all" and 10 for "worst pain possible".
Pre operative pain | Intraoperative
  Pain score at surgical incision (start of surgical procedure) will be assessed via a Numerical Rating Scale (NRS). This scale is ranged (0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10) in which 0 stand for "no pain at all" and 10 for "worst pain possible".
Intra-operative: pain | Intraoperative
  The pain score will be assessed over the period of the surgical procedure (which starts with the incision and ends with the closure of the surgical incision). The pain score will be assessed via a Numerical Rating Scale (NRS). This scale is ranged (0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10) in which 0 stand for "no pain at all" and 10 for "worst pain possible".
Time in operating room | Intraoperative
  Time patient is in operating room
Time of surgical procedure | Intraoperative
  Time of surgical procedure
Post-operative pain | 1 day
  Average pain score at hospital discharge and at day 1 after surgery will be assessed via a Numerical Rating Scale (NRS). This scale is ranged (0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10) in which 0 stand for "no pain at all" and 10 for "worst pain possible".
Use of post-operative pain medication | 1 day
  The use of pain medication after surgery and at day 1 after surgery will be investigated and specified (type, dosage and frequency of medication)
Patient satisfaction | 1 day
  General satisfaction of the patient with the anesthesia technique will be assessed via a 7-point Likert Scale. This scale is ranged (1, 2, 3, 4, 5, 6, 7) in which 1 stands for "completely dissatisfied" and 7 for "completely satisfied".
Surgeon satisfaction | 1 day
  Satisfaction of the surgeon with the surgical conditions will be assessed via a 7-point Likert Scale. This scale is ranged (1, 2, 3, 4, 5, 6, 7) in which 1 stands for "completely dissatisfied" and 7 for "completely satisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Björn Stessel, MD, PhD, Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mariano ER, Lehr MK, Loland VJ, Bishop ML. Choice of loco-regional anesthetic technique affects operating room efficiency for carpal tunnel release. J Anesth. 2013 Aug;27(4):611-4. doi: 10.1007/s00540-013-1578-8. Epub 2013 Mar 5. PMID 23460418
- [Background] Soberon JR Jr, Crookshank JW 3rd, Nossaman BD, Elliott CE, Sisco-Wise LE, Duncan SF. Distal Peripheral Nerve Blocks in the Forearm as an Alternative to Proximal Brachial Plexus Blockade in Patients Undergoing Hand Surgery: A Prospective and Randomized Pilot Study. J Hand Surg Am. 2016 Oct;41(10):969-977. doi: 10.1016/j.jhsa.2016.07.092. Epub 2016 Aug 11. PMID 27524691
- [Derived] Jalil H, Polfliet F, Nijs K, Bruckers L, De Wachter G, Callebaut I, Salimans L, Van de Velde M, Stessel B. Efficacy of ultrasound-guided forearm nerve block versus forearm intravenous regional anaesthesia in patients undergoing carpal tunnel release: A randomized controlled trial. PLoS One. 2021 Feb 19;16(2):e0246863. doi: 10.1371/journal.pone.0246863. eCollection 2021. PMID 33606754